CLINICAL TRIAL: NCT03171480
Title: Randomized Controlled Trial of Nitric-oxide Donor (NOD) Isosorbide Mononitrate (IMN) Versus Placebo for Induction of Labor in Pregnancies Complicated by Preeclampsia
Brief Title: Use of Nitrous Oxide Donor for Labor Induction in Women With PreEclampsia
Acronym: NOPE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kara M Rood, MD, MD, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017H0195
Record Dates: First submitted 2017-05-10; First posted 2017-05-31 (Actual); Results first posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Preeclampsia; Labor, Premature
Keywords: Preeclampsia; Induction
MeSH Terms: conditions — Pre-Eclampsia; Obstetric Labor, Premature | interventions — isosorbide-5-mononitrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A double blinded, placebo controlled, randomized clinical trial of patients undergoing induction of labor for preeclampsia. Study drug or identical appearing placebo will be delivered to labor floor by pharmacist, after randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Monoket pill (Experimental): Isosorbide mononitrate is a drug used principally in the treatment of angina pectoris[1] and acts by dilating the blood vessels so as to reduce the blood pressure. It is sold in the USA by Kremers Urban under the trade name Monoket, also sold in the USA under the name Imdur,
  Interventions: Drug: Monoket Pill
- Placebo pill (Placebo Comparator): The pharmacy has compounded an identical appearing placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Monoket Pill — Intra-vaginal application of Monoket as a cervical ripening agent for pregnant women undergoing induction of labor
  Other Names: Isosorbide mononitrate
  Arms: Monoket pill
Drug: Placebo — The pharmacy has compounded an identical appearing placebo
  Arms: Placebo pill

SUMMARY:
A randomized controlled trial (RCT) of nitric-oxide donor (NOD) isosorbide mononitrate (IMN) versus placebo as an adjuvant to misoprostol/ intra-cervical Foley bulb for induction of labor to decrease rate of cesarean deliveries in pregnancies complicated by preeclampsia (≥24/0 weeks' gestation)

DETAILED DESCRIPTION:
The investigators are proposing a double blinded, placebo controlled, randomized clinical trial of patients undergoing induction of labor for preeclampsia. Once the decision to induce will be taken, the participants will be randomized to receive either intravaginal IMN (40mg) or identical appearing placebo placed every 4hrs in the posterior vaginal fornix X 3 doses. IMN or placebo will be discontinued when active labor occurs or when the physician decides to proceed with augmentation with oxytocin or AROM. Participants will be induced using the investigators routine induction agents, Misoprostol (25 mcg every 4 hrs for maximum of 6 doses) and an intra-cervical foley bulb will be inserted with 2nd dose of IMN or placebo. Regarding management of labor, physician decides when to proceed with augmentation with oxytocin or AROM.

ELIGIBILITY:
Inclusion Criteria:

* Women older than 18 years at the time of induction of labor with the ability to give informed consent
* Induction of labor for clinical diagnosis of preeclampsia
* Unfavorable cervix (Bishop's score of less than 6)
* Cervical dilation 2cm or less
* Singleton
* Gestational age ≥ 24 weeks
* English speaking

Exclusion Criteria:

* • Contraindication to vaginal delivery

  * Contraindication to misoprostol
  * Fetal Demise
  * Major fetal anomaly
  * Non-english speaking women
  * HIV
  * Medical conditions requiring assisted second stage
  * Category III tracing
  * Eclampsia
  * Hemolysis Elevated Liver enzymes Low Platelets syndrome
  * DIC or active hemorrhage before randomization
  * Hypersensitivity to isosorbide mononitrate
  * Isosorbide mononitrate should not be used in cases of acute myocardial infarction with low filling pressure, acute circulatory failure (shock, vascular collapse), or hypertrophic obstructive cardiomyopathy (HOCM), constrictive pericarditis, low cardiac filling pressures, aortic/mitral valve stenosis and diseases associated with a raised intra-cranial pressure e.g following a head trauma and including cerebral hemorrhage.
  * Isosorbide mononitrate should not be used in patients with severe anemia, severe hypotension, closed angle glaucoma or severe hypovolaemia.
  * Isosorbide mononitrate tablets contain lactose and therefore patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption should not take this medicine.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only pregnant women with preeclampsia
Enrollment: 176 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara Rood, MD, Principal Investigator — The Ohio State Wexner Medical Center
Locations (1):
- The Ohio State Medical Center Labor and Delivery Unit, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buhimschi I, Ali M, Jain V, Chwalisz K, Garfield RE. Differential regulation of nitric oxide in the rat uterus and cervix during pregnancy and labour. Hum Reprod. 1996 Aug;11(8):1755-66. doi: 10.1093/oxfordjournals.humrep.a019481. PMID 8921128
- [Background] Ghosh A, Lattey KR, Kelly AJ. Nitric oxide donors for cervical ripening and induction of labour. Cochrane Database Syst Rev. 2016 Dec 5;12(12):CD006901. doi: 10.1002/14651858.CD006901.pub3. PMID 27918616
- [Background] Chanrachakul B, Herabutya Y, Punyavachira P. Randomized trial of isosorbide mononitrate versus misoprostol for cervical ripening at term. Int J Gynaecol Obstet. 2002 Aug;78(2):139-45. doi: 10.1016/s0020-7292(02)00128-5. PMID 12175715
- [Background] El-Khayat W, Alelaiw H, El-kateb A, Elsemary A. Comparing vaginal misoprostol versus Foley catheter plus vaginal isosorbide mononitrate for labor induction. J Matern Fetal Neonatal Med. 2016;29(3):487-92. doi: 10.3109/14767058.2015.1007036. Epub 2015 Feb 19. PMID 25694257
- [Background] Thomson AJ, Lunan CB, Cameron AD, Cameron IT, Greer IA, Norman JE. Nitric oxide donors induce ripening of the human uterine cervix: a randomised controlled trial. Br J Obstet Gynaecol. 1997 Sep;104(9):1054-7. doi: 10.1111/j.1471-0528.1997.tb12066.x. PMID 9307534
- [Result] Collingham JP, Fuh KC, Caughey AB, Pullen KM, Lyell DJ, El-Sayed YY. Oral misoprostol and vaginal isosorbide mononitrate for labor induction: a randomized controlled trial. Obstet Gynecol. 2010 Jul;116(1):121-126. doi: 10.1097/AOG.0b013e3181e408f2. PMID 20567177
- [Derived] Gee SE, Ma'ayeh M, Cackovic H, Samuels P, Thung SF, Landon MB, Rood KM. Addition of vaginal isosorbide mononitrate for labor induction in pregnancies complicated by hypertensive diseases of pregnancy: a randomized controlled trial. Am J Obstet Gynecol MFM. 2021 Jul;3(4):100343. doi: 10.1016/j.ajogmf.2021.100343. Epub 2021 Feb 27. PMID 33652160

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: The pharmacy has compounded an identical appearing placebo
  Monoket Pill: Intra-vaginal application of Monoket as a cervical ripening agent for pregnant women undergoing induction of labor
Period: Overall Study
Arm/Group | Monoket Pill | Placebo
Started | 89 | 87
Completed | 89 | 87
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Pill: The pharmacy has compounded an identical appearing placebo
  Monoket Pill: Intra-vaginal application of Monoket as a cervical ripening agent for pregnant women undergoing induction of labor
- Total: Total of all reporting groups
Arm/Group | Monoket Pill | Placebo Pill | Total
Number analyzed (Participants) | 89 | 87 | 176
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 89 | 87 | 176
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 28 [23 to 32] | 27 [23 to 31] | 28 [23 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 87 | 176
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Cesarean Delivery Rate
Description: Rate of cesarean section for those enrolled in study
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Monoket Pill | Placebo
Number analyzed (Participants) | 89 | 87
Participants | 29 | 22

2. Secondary Outcome: Placental Abruption, Use of IV Antihypertensive Drug, Maternal Hypotension, Uterine Hyperstimulation and Meconium Stained Fluid
Description: placenta abruption at time of delivery, administration of IV antihypertensive medication for BP >160/110, maternal hypotensive defined as <90/50, Uterine hyperstimulation defined as >3 contractions in 10 minutes and meconium stained amniotic fluid anytime during labor induction/augmentation
Time Frame: during the induction of labor till delivery for all outcomes
Measure: Count of Participants; unit: Participants
Arm/Group | Monoket Pill | Placebo Pill
Number analyzed (Participants) | 89 | 87
Participants
  Abruption | 0 | 0
  Anti-hypertensives | 29 | 32
  hypotension | 9 | 8
  uterine hyperstimulation | 3 | 1
  MSAF | 0 | 0

ADVERSE EVENTS:
Time Frame: During hospitalization for delivery
Description: Adverse event was defined as unexpected and unanticipated side effect form administration of the medication (IMN)
Arm/Group | Monoket Pill | Placebo
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/87
Other Adverse Events (participants affected / at risk) | 0/89 | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT03171480/Prot_SAP_000.pdf